CLINICAL TRIAL: NCT05015972
Title: A Study of CTA30X UCAR-T Cell Injection in the Treatment of Patients With r/r CD19+ B Hematologic Malignancies
Brief Title: UCAR-T for CD19+ Refractory/Relapsed B Hematologic Malignancies
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: No proper participant is found.
Sponsor: 920th Hospital of Joint Logistics Support Force of People's Liberation Army of China (Other)
Collaborators: Nanjing Bioheng Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTA30X
Record Dates: First submitted 2021-04-21; First posted 2021-08-23 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: B-cell Lymphoma
Keywords: UCAR-T; allogeneic; CD19; B-ALL; B-NHL
MeSH Terms: conditions — Lymphoma, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CTA30X UCAR-T treatment (Experimental): CD19+ R/R B Hematologic Malignancies patients be treated with a single dose of CTA30X UCAR-T cells. Total dose of(5-30)*10E6/kg cells will be administered at Day 0
  Interventions: Biological: CTA30X UCAR-T injection

INTERVENTIONS:
Biological: CTA30X UCAR-T injection — CTA30X UCAR-T injection is an allogeneic CAR-Ttargeted CD19 . A single infusion of CART cells will be administered intravenously.

SUMMARY:
This is a single arm, open-label, single-center prospective study to determinethe safety and efficacy of CTA30X UCAR-T cells in patients diagnosed with CD19+ refractory/relapsed B Hematologic Malignancies

DETAILED DESCRIPTION:
The main aim of the study is to determine the safety and efficacy of CTA30X UCAR-T in R/R B Hematologic Malignancies. CTA30X UCAR-T is an allogeneic chimeric antigenreceptor T-cell (CAR-T) therapy that targets CD19 and B-cell Hematologic Malignancies. The study will include 72 subjects to receive CTA30X UCAR-T singleinfusion.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria applicable only to ALL:

1. Age ≥3 and < 70 years old, gender is not limited;
2. Patients with a histologic diagnosis of CD19+ B-ALL according to the National Comprehensive Cancer Network (NCCN) Clinical Practice Guidelines for Acute Lymphoblastic Leukemia (2016.v1);
3. Meet the R/R CD19+ B-ALL diagnosis, including any of the following conditions:

   A) No CR after standard chemotherapy; B) CR was induced for the first time, but the duration of CR was less than 12 months; C) R/R CD19+ B-ALL that failed after the first or repeated remedial therapy; D) 2 or more recurrences;
4. Number of primary cells (primary + juvenile) in bone marrow, > 5% (morphology) and/or > 1% (flow cytometry);
5. Philadelphia chromosomal negative (PH -) subjects;Philadelphia chromosomal positive (pH +) subjects who either cannot tolerate or do not respond to either of the TKI treatments;

Inclusion criteria for NHL only:

1. Age ≥18 years old and < 70 years old, regardless of gender;
2. According to the 2016 WHO classification criteria for lymphocytic tumors, the histological diagnosis included: DLBCL (NOS);Subjects with follicular lymphoma, chronic lymphocytic leukemia/small lymphocytic lymphoma transformation, and PMBCL and high-grade B-cell lymphoma;
3. Relapsed or refractory B-NHL (meets one of the following conditions) :

   A) Subjects have no remission or recurrence after receiving second-line chemotherapy regimen or above; B) primary drug resistance; C) Subjects relapse after autologous hematopoietic stem cell transplantation;
4. According to Lugano 2014 criteria, there should be at least one evaluable tumor focus;

Common standards for ALL and NHL:

1. Serum total bilirubin ≤51 umol/L, serum ALT and AST ≤ 3 times of the upper limit of the normal range, serum creatinine ≤176.8 umol /L;
2. Echocardiography showed left ventricular ejection fraction (LVEF) ≥50%;
3. Subjects have no active pulmonary infection, and oxygen saturation of suction finger vein is ≥92%;
4. The estimated survival time is more than 3 months;
5. ECOG score 0-2;
6. Subjects or their legal guardians participate in this study voluntarily and sign the informed consent.

Exclusion Criteria:

1. Extramedullary lesions, except those with effectively controlled CNSL (CNS-1);(All patients only)
2. A lymphoblastic crisis of chronic myeloid leukemia, Burkitt's leukemia/lymphoma, was diagnosed according to WHO classification;(All patients only)
3. having a genetic syndrome such as Fanconi anemia, Kostmann syndrome, Shwachman syndrome or any other known bone marrow failure syndrome;(All patients only)
4. Extranodal intracranial lesions (tumor cells in CSF and/or intracranial lymphoma shown on MRI);(For patients with NHL only)
5. subjects with extensive gastrointestinal lymphoma invasion;(For patients with NHL only)
6. Subjects received radiotherapy, chemotherapy and monoclonal antibody treatment within 1 week before screening;
7. Have a history of allergy to any one ingredient in cell products;
8. Prior use of any CAR T cell product or other genetically modified T cell therapy
9. Subjects with cardiac dysfunction grade III or IV according to the New York Heart Association (NYHA) cardiac function classification standards;
10. Myocardial infarction, cardiac angioplasty or stenting, unstable angina pectoris or other clinically serious heart disease within 12 months of enrollment;
11. Severe primary or secondary hypertension of grade 3 or higher (WHO Hypertension Guidelines, 1999);
12. Patients with prolonged QT interval indicated by ECG and previous severe heart disease such as severe arrhythmia;
13. Previous history of craniocerebral trauma, disturbance of consciousness, epilepsy, cerebrovascular ischemia, cerebrovascular hemorrhagic disease, etc.
14. Severe active infection (except simple urinary tract infection and bacterial pharyngitis);
15. Subject has a history of other primary cancers except for:

    A. Non-melanoma cured by excision, such as basal cell carcinoma of the skin; B. Cervical carcinoma in situ, local prostate cancer, and ductal carcinoma in situ with disease-free survival ≥2 years after adequate treatment;
16. Subjects with autoimmune diseases requiring treatment or subjects requiring immunosuppressive therapy;
17. Patients with graft-versus-host disease (GVHD) and/or requiring immunosuppressive therapy;
18. Live vaccine inoculation within 4 weeks before screening;
19. Subjects have a history of alcohol, drug abuse or mental illness;
20. During screening, if the subjects were HBV surface antigen positive, they were tested by active hepatitis B PCR. If HBV DNA copy number > 1000, they were excluded; if HBV DNA copy number ≤1000, routine antiviral treatment was required after enlistment).Hepatitis C, syphilis antibody positive, syphilis virus DNA test exceeded the upper limit of normal value and CMV virus DNA test exceeded the upper limit of normal value;
21. Subjects who were receiving systemic steroid therapy prior to screening and were determined by the investigator to require long-term systemic steroid therapy during the treatment period (other than inhalation or topical use);
22. Screening participants who had participated in other clinical trials within the previous 2 weeks;
23. Pregnant and lactating women and fertile subjects who are unable to take effective contraceptive measures (both male and female);
24. Any situation that the investigator believes may increase the risk to the subject or interfere with the outcome of the study.

Ages: 3 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-08-20 (Estimated); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity | Up to 24 weeks after CAR-T infusion
  CRS lasting ≥7 days G3 or ≥G4 after CTA30X infusion;
Incidence of AE after CAR-T infusion | Up to 4 weeks after the infusion of CAR-T cells
  Incidence of adverse events after CTA30X UCAR-T infusion

SECONDARY OUTCOMES:
ORR rate | 1month, 3months after CTA30X UCAR-T infusion
  Overall response rate (ORR=CR+CRi) after CTA30X UCAR-T infusion
MRD-ORR | within 3months after CTA30X UCAR-T infusion
  The overall response rate was MRD negative within 3 months after treatment
BOR | within 3months after CTA30X UCAR-T infusion
  The best overall response within 3 months after treatment
DOR | From the onset of a tumor from the first assessment of CR or PR up to 1 year
  Duration of remission
ORR | 6month, 12months、 18months and24months after CTA30X UCAR-T infusion
  ORR=CR+CRi
EFS | 6month, 12months、 18months and24months after CTA30X UCAR-T infusion
  Event-free survival
OS | 6month, 12months、 18months and24months after CTA30X UCAR-T infusion
  Overall survival

OTHER OUTCOMES:
exploratory | up to 24 months after CAR-T infusion
  The proliferation and survival time of CAR T cells in vivo and the clearance rate of B cells.

CONTACTS AND LOCATIONS:
Locations (1):
- No.212 Daguan Road, Xishan District, Kunming, Yunnan, China